CLINICAL TRIAL: NCT02447679
Title: Oral Thalidomide and Tegafur-uracil to Decrease Hepatocellular Carcinoma Recurrent After Hepatectomy in High Risk Patients -A Phase II Study
Brief Title: Oral Thalidomide and Tegafur-uracil to Decrease Hepatocellular Carcinoma Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CGMF-IRB-97-1291A
Record Dates: First submitted 2014-12-16; First posted 2015-05-19 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-12

CONDITIONS: Adult Hepatocellular Carcinoma; Recurrent Hepatocellular Carcinoma; Adverse Reaction to Drug; Vascular Endothelial Growth Factor Overexpression
MeSH Terms: conditions — Carcinoma, Hepatocellular; Drug-Related Side Effects and Adverse Reactions | interventions — Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- thalidomine (Experimental): 1. Thalidomide 400mg/day for 1 year
  2. tegafur-uracil 2 tables for 1 year.
  Interventions: Drug: thalidomine; Drug: tegafur-uracil

INTERVENTIONS:
Drug: thalidomine — thalidomine (400mg/day) for 1 year to prevent HCC recurrence
  Other Names: thado
Drug: tegafur-uracil — tegafur-uracil (2 tablelet twice a day) for 1 year to prevent HCC recurrence
  Other Names: ufur

SUMMARY:
This single-centered phase II clinical study is to obtain preliminary information on 1-year recurrence-free survival rate, recurrence-free survival and safety profile of thalidomide in combination with tegafur-uracil in hepatocellular carcinoma after hepatectomy and explore biomarkers(VEGF/bFGF) for thalidomide response.

DETAILED DESCRIPTION:
After liver resection to remove the hepatocellular carcinioma completely, the patients with high risk of tumor recurrence will be enrolled into this study. The high risk of tumor recurrence depends on tumor characteristics. The risk factors of tumor characteristics included tumor size >5 cm in diameter, abscence of encapsulation, vascular invasion and presence of daughter nodules. The patients with high risk of tumor recurrence will have 1 to 3 risk factors. When the patients are enrolled into the study, oral thalidomide in combination with tegafur-uracil will be applied to prevent tumor recurrence. The patients will be fillowed uo erevy 3 mnoths.

ELIGIBILITY:
Inclusion Criteria:

1. stage I-III（TNM: T1-T3） hepatocellular carcinoma
2. previously received curative surgery
3. presence at least one and no more than three of the following risk factors ,

i.Tumor size ≧ 5 cm ii.presence of microscopic or macrovascular venous invasion iii.presence of satellite nodules/addition nodules iv.no capsular formation v.multiple tumors d.performance status of ECOG 0, 1 e.age between 20 and 75 years f.no residual or recurrent tumors detected by computed tomography (CT) or echo within 3-6 weeks after surgery g.written informed consent to participate in the trial

Exclusion Criteria:

1. other malignancy with the exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ prior to the entry of study
2. previously received chemotherapy
3. less than 2 weeks since previous radiotherapy/surgery
4. white blood cell (WBC) less than 3,000/mm3 and absolute neutrophil count (ANC) less than 1,500/mm3, and platelets less than 100,000/mm3
5. serum bilirubin greater than 1.5 times the upper limit of normal range (ULN)
6. alanine aminotransferase (ALT) or aspartate transaminase (AST) greater than 5 times the ULN
7. alkaline phosphatase greater than 5 times the ULN
8. presence of serious concomitant illness which might be aggravated by study medication:uncontrolled infection (active serious infections that are not controlled by antibiotics)
9. hypersensitivity to thalidomide or compounds pregnant or breast feeding women, or women of child-bearing potential unless using two reliable and appropriate contraceptive method

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
tumor recurrence | every 3 months, up to 5 years
  Measure a-fetoprotein and perform liver echo to find out tumor recurrence every 3 month. Then, if a tumor/tumors are found in liver echo, tumor recurrence will be confirmed by CT scan. The imaging on CT shows typical HCC pattern.
  The pilot study is to obtain preliminary information on:
  * 3-year recurrence-free survival rate
  * Recurrence-free survival
  * Safety profile of the treatment
  * Biomarkers response(VEGF/bFGF)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Lee, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan